CLINICAL TRIAL: NCT05441800
Title: Epidemiology and Clinical Characteristics of Emerging and Re-emerging Infectious Diseases
Brief Title: Epidemiology and Clinical Characteristics of Emerging and Re-emerging Infectious Diseases With Epidemic Potential in Mali
Acronym: ECERID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Clinical Research Center, Mali (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: UCRC-001
Record Dates: First submitted 2022-06-07; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Febrile Illness
Keywords: Unknown febrile; emerging or; re-emerging infectious disease
MeSH Terms: conditions — Communicable Diseases, Emerging | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Blood samples, Other samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Study — observational study to include participants with a spectrum of emerging or unknown pathogens with the objective to determine etiology and clinical characteristics of those diseases

SUMMARY:
This is a prospective observational study to include participants with a spectrum of emerging or unknown pathogens with the objective to determine etiology and clinical characteristics of those diseases.

DETAILED DESCRIPTION:
Infectious diseases remain one of the leading causes of death worldwide despite innovations in medical research and the availability of new treatments. Emerging diseases include outbreaks of previously unknown diseases or known diseases where the incidence in humans has significantly increased in the past two decades. Detailed studies on emerging and re-emerging infectious agents to better understand pathogens' biology and host pathogenesis are mostly lacking. This study protocol is to prepare for a rapid coordinated clinical investigation of acute infections of emerging and re-emerging infectious agents in Mali. In collaboration with the Mali Ministry of Health and Public Hygiene, we will conduct an observational study to include participants with a spectrum of emerging or unknown pathogens with the objective to determine etiology and clinical characteristics of those diseases. Patients with suspected emerging or re-emerging infectious diseases within 15 km of Point G Hospital in Bamako will be invited to participate in this study.

ELIGIBILITY:
Participants referred or managed by the National Disease Surveillance Committee, primary healthcare facilities, level-3 hospitals, or other facilities Adults and children of any age

Unexplained fever (temperature greater than or equal to 38°C), recorded or reported, within 24 to 48 hours, regardless duration with at least one of the following signs or symptoms:

* Unexplained bleeding
* One or more generic symptoms (headache, tiredness, myalgia, arthralgia, diarrhea, anorexia, weight loss, rash)
* Jaundice
* One or more respiratory symptoms (cough, dyspnea, pharyngitis, rhinorrhea)
* Guillain-Barré syndrome
* Newborns with microcephaly or other brain defects
* Agree to have samples collected and stored for further studies

Exclusion criteria

- Participants may be excluded from enrolling in the study if they have any known medical disorders or other circumstances which, in the opinion of the investigator, might make participation unsafe or difficult (e.g. inability to obtain necessary samples, mental illness).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects enrolled in this study will be identified by the National Epidemiological Monitoring Committee, the Department of Infectious and Tropical Diseases, or other services of the level-3 hospitals in the context of public health emergency or epidemic. Participants will be suspected of having a febrile illness due to an infectious pathogen that has not been formally identified by existing diagnostic strategies or standard of care testing.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-06-18 (Estimated); Study Completion 2023-06-18 (Estimated)

PRIMARY OUTCOMES:
Identify the etiologies and immediate outcomes of emerging and re-emerging diseases in Mali. | In 3 years
  To identify the etiologies (e.g. lassa fever, measles, covid-19, zika, Ebola virus disease) of unexplained febrile illnesses in adults and children in Mali measured by the proportion of cases identified who are children, or who are adults.

CONTACTS AND LOCATIONS:
Overall Officials: Sounkalo DAO, MD, Principal Investigator — University of Science, Techniques and Technologies of Bamako, Mali
Locations (1):
- University Clinical Research Center (UCRC) / USTTB, Bamako, Mali